CLINICAL TRIAL: NCT02331550
Title: Observational vs. Ablative Treatment for Low-grade Squamous Intraepithelial Lesions. Retrospective Paired Cohort Study.
Brief Title: Observational vs. Ablative Treatment for Low-grade Squamous Intraepithelial Lesions.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Thomas Hospital, Panama (Other)
Responsible Party: Principal Investigator, Osvaldo A. Reyes T., Coordinator of Research, Saint Thomas Hospital, Panama
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MHST2014-01
Record Dates: First submitted 2015-01-03; First posted 2015-01-06 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: LSIL, Low-Grade Squamous Intraepithelial Lesions
Keywords: Low-Grade Squamous Intraepithelial Lesions
MeSH Terms: conditions — Squamous Intraepithelial Lesions | interventions — Watchful Waiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Expectant treatment (Experimental): Patients diagnosed with Low-Grade Squamous Intraepithelial Lesions that were managed with observation and evaluation at 6 and 12 months after diagnosis.
  Interventions: Procedure: Expectant management
- Ablative treatment (Experimental): Patients diagnosed with Low-Grade Squamous Intraepithelial Lesions that were managed with an ablative treatment and evaluated at 6 and 12 months after diagnosis.
  Interventions: Procedure: Ablative treatment

INTERVENTIONS:
Procedure: Ablative treatment — Use of an ablative treatment (cryotherapy) for the management of Low-Grade Squamous Intraepithelial Lesions of the cervix.
  Arms: Ablative treatment
Procedure: Expectant management — Patients diagnosed with Low-Grade Squamous Intraepithelial Lesions were managed with observation and evaluation at 6 and 12 months after diagnosis.
  Arms: Expectant treatment

SUMMARY:
To evaluate the rate of regression and progression of low-grade squamous intraepithelial lesion comparing expectant vs. ablative treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Low-Grade Squamous Intraepithelial Lesion by cervical cytology.
* Positive Biopsy for Low-Grade Squamous Intraepithelial Lesion after colposcopy.

Exclusion Criteria:

* Serological detection of human immunodeficiency virus (HIV).

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2014-01; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Number of patients diagnosed with Low-Grade Squamous Intraepithelial Lesions that progressed to a higher level lesion (High Grade or cervical cancer) when evaluated at 6 and 12 months after diagnosis. | 12 months

SECONDARY OUTCOMES:
Number of patients diagnosed with Low-Grade Squamous Intraepithelial Lesions that regressed to a higher level lesion (High Grade or cervical cancer) when evaluated at 6 and 12 months after diagnosis. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Osvaldo Reyes, MD, Principal Investigator — Saint Thomas Hospital, Panama
Locations (1):
- Saint Thomas H, Panama City, Provincia de Panamá, Panama